CLINICAL TRIAL: NCT05720026
Title: A Multicenter, Randomized, Double-Blind, Parallel-Controlled Phase Ⅲ Clinical Study to Compare the Efficacy and Safety of SYSA1901 vs Pertuzumab (Perjeta®) in the Neoadjuvant Therapy of HER2-Positive Breast Cancer
Brief Title: Study to Evaluate the Efficacy and Safety of SYSA1901 vs. Perjeta® of HER2-Positive Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSA1901-002
Record Dates: First submitted 2022-11-25; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pertuzumab; Trastuzumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): SYSA1901 combined with trastuzumab and docetaxel will be administrated intravenously on a 3-weekly schedule for 4 cycles (21 days per cycle).
  Interventions: Drug: SYSA1901; Drug: Trastuzumab; Drug: Docetaxel
- Control group (Active Comparator): Perjeta® combined with trastuzumab and docetaxel will be administrated intravenously on a 3-weekly schedule for 4 cycles (21 days per cycle).
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: SYSA1901 — loading dose of 840 mg IV, followed by 420 mg IV, q3w/cycle, total 4cycle
  Other Names: pertuzumab biosimilar
  Arms: Treatment group
Drug: Pertuzumab — loading dose of 840 mg IV, followed by 420 mg IV, q3w/cycle, total 4cycle
  Other Names: Perjeta®
  Arms: Control group
Drug: Trastuzumab — loading dose of 8 mg/kg IV, followed by 6 mg/kg IV, q3w/cycle, total 4cycle
  Other Names: Herceptin®
Drug: Docetaxel — 75 mg/m^2 IV, q3w/cycle, total 4cycle
  Other Names: Docetaxel injection

SUMMARY:
This is a phase Ⅲ, double-blind, randomized, parallel-controlled, multicenter equivalence study to compare the efficacy and safety of SYSA1901 + trastuzumab + docetaxel vs. Perjeta® + trastuzumab + docetaxel in the participants with early-stage or locally advanced HER2-positive and HR-negative breast cancer with a primary tumor > 2 cm.

DETAILED DESCRIPTION:
This is a phase Ⅲ, double-blind, randomized, parallel-controlled, multicenter equivalence study to compare the efficacy and safety of SYSA1901 + trastuzumab + docetaxel vs. Perjeta® + trastuzumab + docetaxel in the patients with early-stage or locally advanced HER2-positive and HR-negative breast cancer with a primary tumor > 2 cm. The eligible patients will be randomized to treatment group (SYSA1901 + Trastuzumab + Docetaxel) or control group (Perjeta® + Trastuzumab + Docetaxel) at 1:1 ratio. The stratification factor is disease category (early-stage vs. locally advanced).

The primary endpoint is total pCR (tpCR). Secondary efficacy endpoints include breast pCR (bpCR), objective response rate (ORR)，pharmacokinetic (PK) and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent;
2. Age ≥ 18 years;
3. Histologically confirmed invasive breast carcinoma, and breast cancer staging [in accordance with the American Joint Committee on Cancer (AJCC) staging system (8th edition)]: early-stage (T2-3, N0-1, M0) or locally advanced (T2-3, N2-3, M0; T4, any N, M0);
4. Eastern Cooperative Oncology Group (ECOG) performance status: 0-1;
5. HER2 positive, defined as immunohistochemistry (IHC) 3+, or IHC 2+ with In Situ Hybridization (ISH) positive;
6. Estrogen receptor (ER) and progestin receptor (PR) negative; ER and PR negative is defined as < 1% nuclear staining;
7. Agree to receive surgical treatment of breast cancer at the participating unit when the surgical criteria are met after neoadjuvant therapy;
8. Primary tumor size of > 2 cm in diameter;
9. Left ventricular ejection fraction (LVEF)≥ 55% measured by echocardiography (ECHO) or multiple gated acquisition (MUGA) scan;
10. Adequate major organ function, meeting the following criteria (have not received blood transfusion, EPO,G-CSF, other hematopoietic stimulating factors or medical supportive treatments within 14 days before the first dose of study drug): absolute neutrophil count (ANC) ≥1.5×10^9 /L; Leukocyte count≥3.0×10^9 /L, platelet (PLT) ≥100×10^9 /L; hemoglobin ≥90 g/L; Serum creatinine ≤ 1.5 x the upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; total bilirubin ≤1.5×ULN; international normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN, or activated partial thromboplastin time (APTT) ≤1.5×ULN (not receiving anticoagulation), or patients receiving anticoagulation need to be within treatment target range and at a stable dose;
11. Women of childbearing age must have a negative pregnancy test prior to the first dose;
12. Female and male patient of childbearing age must agree to take adequate contraceptive measures during the entire study period and through at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer, inflammatory breast cancer, and bilateral breast cancer;
2. Previous severe allergic reactions to any drug or its components in this trial (NCI-CTCAE 5.0 grade greater than 3);
3. Patients with any other malignant tumor within 2 years (except for skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, local prostate cancer, in situ cervical cancer and other malignant tumors that have been radically removed and have not recurred);
4. Major surgery and incomplete recovery within 4 weeks prior to the first dose of study drug;
5. Patients have received other clinical trial drugs within 4 weeks before the first dose of study drug;
6. Received chemotherapy, endocrine therapy, anti-HER2 biological therapy, breast surgery or local radiotherapy for breast cancer (except for diagnostic biopsy surgery or benign breast tumor surgery);
7. History of immunodeficiency diseases, including human immunodeficiency virus (HIV) positive, active syphilis;
8. History of severe cardiovascular disease, including previous coronary artery bypass grafting or coronary stent implantation, myocardial infarction or cerebrovascular accident within 6 months, history of congestive heart failure or unstable angina pectoris, uncontrolled severe hypertension and arrhythmia requiring drug treatment;
9. Any uncontrollable complication, infection, or other condition that may affect study compliance or interfere with efficacy evaluation;
10. History of drug abuse, or alcoholism, drug addicts;
11. History of neurological or psychiatric disorders and poor compliance, such as epilepsy and dementia;
12. Pregnant and breastfeeding women;
13. Other conditions that may affect the assessment of the primary endpoint or render the patient inappropriate for entry into this study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Total pathologic complete response (tpCR) assessed by Independent Review Committee（IRC） | Up to 5 months
  The tpCR is defined as the histological evidence of no malignancy of lymph nodes in the regions of primary lesion and metastasis of breast cancer (i.e., ypT0/is, ypN0 in accordance with the AJCC staging system)

SECONDARY OUTCOMES:
Percentage of patients with tpCR as assessed by the investigator | Up to 5 months
  The tpCR is defined as the histological evidence of no malignancy of lymph nodes in the regions of primary lesion and metastasis of breast cancer (i.e., ypT0/is, ypN0 in accordance with the AJCC staging system)
Breast pathologic complete response (bpCR) assessed by IRC | Up to 5 months
  The bpCR is defined as the histological evidence of no malignancy in the primary lesion of breast cancer, or only carcinoma in situ (i.e., ypT0/Tis, in accordance with current AJCC staging system).
Breast pathologic complete response (bpCR) assessed by the investigator | Up to 5 months
  The bpCR is defined as the histological evidence of no malignancy in the primary lesion of breast cancer, or only carcinoma in situ (i.e., ypT0/Tis, in accordance with current AJCC staging system).
Percentage of patients with an objective response (BORR) | Prior to surgery
  An objective response is defined as the percentage of patients who achieved a complete response or partial response as the best tumor response during the treatment period (that is, during Cycles 1-4 prior to surgery), as determined by the investigator on the basis of Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Incidence of adverse event | Up to approximately 30 months after randomization
  Including type, incidence, severity, time and so on of adverse events
Pharmacokinetic parameters of SYSA1901 | Up to approximately 30 months after randomization
  To measure the serum concentration of SYSA1901 and pertuzumab (Perjeta ®) .
Immunogenicity of SYSA1901 | Up to approximately 30 months after randomization
  Anti-drug antibody (ADA) and neutralizing antibody (Nab) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Shao Zhimin, Professor, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China